CLINICAL TRIAL: NCT02634320
Title: Safety and Tolerability of Initiating Aripiprazole Lauroxil in Subjects With Schizophrenia Who Are Inadequately Treated With Paliperidone Palmitate or Risperidone Long Acting Injection
Brief Title: A Study of Aripiprazole Lauroxil (Also Known as ARISTADA TM) in Subjects With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALK9072-A401
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Results first posted 2018-11-08 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Schizophrenia
Keywords: Alkermes; ARISTADA; Aripiprazole Lauroxil; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — aripiprazole lauroxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aripiprazole Lauroxil (Other): Intramuscular (IM) injection
  Interventions: Drug: Aripiprazole Lauroxil

INTERVENTIONS:
Drug: Aripiprazole Lauroxil — Monthly IM injection
  Other Names: ARISTADA

SUMMARY:
This study will evaluate the safety and tolerability of aripiprazole lauroxil (also known as ARISTADA, ALKS 9070).

ELIGIBILITY:
Inclusion Criteria:

* Has demonstrated tolerability to test doses of oral aripiprazole during screening; OR has a history of tolerated use of aripiprazole
* Has a diagnosis of schizophrenia
* Is clinically stable
* Has received at least 3 doses of risperidone long acting injection (Risperdal Consta) or paliperidone palmitate (Invega Sustenna) prior to screening.
* Has no antipsychotic medication regimen change for 4 weeks prior to Day 1
* Agreed to abide by the contraceptive requirements o the protocol
* Resides in a stable living situation
* Additional criteria may apply

Exclusion Criteria:

* Is currently pregnant or breastfeeding, or is planning to become pregnant during the study
* Has received Invega Trinza, aripiprazole lauroxil, or IM depot aripiprazole within 6 months of screening
* Has participated in a clinical trial involving any investigational product within the past 3 months, or is currently participating in a clinical trial involving an investigational product
* Has a positive urine drug test for illicit use of amphetamines, barbiturates, cocaine, methadone, opiates, phencyclidine at screening
* Additional criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-12; Primary Completion 2017-07-11 (Actual); Study Completion 2017-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Pathak, MD, Study Director — Alkermes, Inc.
Locations (17):
- United States (17):
  - Alkermes Investigational Site, Little Rock, Arkansas
  - Alkermes Investigational Site, Rogers, Arkansas
  - Alkermes Investigational Site, Anaheim, California
  - Alkermes Investigational Site, Culver City, California
  - Alkermes Investigational Site, Garden Grove, California
  - Alkermes Investigational Site, National City, California
  - Alkermes Investigational Site, Oceanside, California
  - Alkermes Investigational Site, Orange, California
  - Alkermes Investigational Site, Panorama City, California
  - Alkermes Investigational Site, Augusta, Georgia
  - Alkermes Investigational Site, Chicago, Illinois
  - Alkermes Investigational Site, Shreveport, Louisiana
  - Alkermes Investigational Site, St Louis, Missouri
  - Alkermes Investigational Site, Garfield Heights, Ohio
  - Alkermes Investigational Site, Lincoln, Rhode Island
  - Alkermes Investigational Site, Dallas, Texas
  - Alkermes Investigational Site, DeSoto, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Opler MGA, Claxton A, McGrory J, Gasper S, Wang M, Yagoda S. Functioning and Cognition in Patients with Schizophrenia After Initiating Treatment with Aripiprazole Lauroxil: Secondary Outcomes and Post Hoc Analysis. Innov Clin Neurosci. 2024 Mar 1;21(1-3):43-51. eCollection 2024 Jan-Mar. PMID 38495608

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects had schizophrenia, and had been taking paliperidone palmitate (PP) or Risperidone long-acting injection (RLAI) with inadequate results for at least 3 doses prior to screening.
Pre-assignment Details: All subjects received 4 to 6 doses of aripiprazole lauroxil in monthly or 6-week intervals.
Period: Overall Study
Arm/Group | Aripiprazole Lauroxil
Started | 51
Completed | 35
Not Completed | 16
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 3
Not completed — Moved out of area | 2
Not completed — Out of window for study visits | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 5
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Population: The Safety population included all subjects who received at least one dose of study drug. All analyses were performed on the Safety population.
Arm/Group | Aripiprazole Lauroxil
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 51
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 25
  White | 22
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Last Treatment Visit in Clinical Global Impressions-Severity (CGI-S) Scores
Description: The CGI-S is a 7-point scale that requires the clinician to assess how mentally ill the patient is in a specific point in time. Results indicate participants evaluated at one of the following categories: "1: normal, not at all ill"; "2: borderline mentally ill"; "3: mildly ill"; "4: moderately ill"; "5: markedly ill"; "6: severely ill"; and "7: among the most extremely ill patients". Results indicate a change in CGI-S score from baseline to last visit in the treatment period based on the observed data.
Time Frame: Up to 7 months
Population: Safety population includes all subjects who received at least 1 dose of study drug and had a last on-treatment visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole Lauroxil
Number analyzed (Participants) | 49
units on a scale | -0.2 (0.87)
Statistical Analysis 1: Comparison: Aripiprazole Lauroxil; Test type: Other — Statistical test is to confirm the change from baseline is statistically different from 0; p = 0.078, t-test, 2 sided — Change from baseline at last on-treatment visit

2. Secondary Outcome: Change From Baseline to Last Treatment Visit in Brief Psychiatric Rating Scale (BPRS) Scores
Description: The BPRS is an instrument for evaluating change in psychopathology in patients with schizophrenia. It consists of 18 items in which clinicians rate patient symptoms on a 7-point scale (1=not present, 7=extremely severe). Scores range from 18 to 126, with higher scores indicative of more severe psychopathology).
Time Frame: Up to 7 months
Population: Safety population includes all subjects who received at least 1 dose of study drug and had a last on-treatment visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole Lauroxil
Number analyzed (Participants) | 49
units on a scale | -2.7 (9.21)

3. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: Up to 7 months
Population: Safety population includes all subjects who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Aripiprazole Lauroxil
Number analyzed (Participants) | 51
Participants | 21

4. Secondary Outcome: Daily and Social Functioning Will be Measured Using the Heinrichs-Carpenter Quality of Life Scale (QLS)
Description: The QLS is a clinician-rated scale that is used to assess health-related quality of life and functioning in patients with schizoprehnia during the preceding 4 weeks. The QLS consists of 21 items in 4 major domains (Intrapsychic Foundations, Interpersonal Relations, Instrumental Role, and Common Objects and Activities). Following a semi-structured interview, each item is rated on a 7-point scale, from 0 (severe impairment) to 6 (normal or unimpaired functioning).
Time Frame: Up to 7 months
Population: Subjects who had at least one dose of study drug and had a last on-treatment visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole Lauroxil
Number analyzed (Participants) | 49
units on a scale | 0.4 (13.11)

5. Secondary Outcome: Characterization of Healthcare Burden Will be Measured Using the Treatment Services Review, Version 6-Modified for Mental Health (mTSR-6)
Description: Responses to 4 mTSR-6 questions have been provided. Results include the number of participants who responded positively to the category during the entire post-baseline treatment period.
Time Frame: Up to 7 months
Measure: Number; unit: participants
Arm/Group | Aripiprazole Lauroxil
Number analyzed (Participants) | 51
participants
  Spent at least 1 overnight as an inpatient | 3
  Attended an outpatient visit for mental health | 17
  Had at least 1 visit to an ER | 6
  Were arrested, picked up, or transported by police | 2

6. Secondary Outcome: Characterization of Family Burden Will be Measured Using the Burden Assessment Scale (BAS)
Description: The BAS is a 19-item scale completed by the caregiver that focuses on specific subjective and objective consequences of families caring for individuals with severe mental disorders. Respondents are required to indicate whether they have experienced each of the types of burden - 'Not at all', 'A little', 'Some' or "A lot' - in the previous four weeks. These are scored 1, 2, 3 and 4, respectively. The total score ranges between 19 and 76. A higher score indicates more perceived burden. Subjects required a reliable informant (caregiver) in order to participate in the study. These caregivers did not receive study treatment, and they are not represented elsewhere in the results data. The data provided indicates the change from baseline to the last treatment visit.
Time Frame: Up to 7 months
Population: Subjects who received at least one dose of study drug, had a last on-treatment visit, and had an unpaid caregiver providing information.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole Lauroxil
Number analyzed (Participants) | 19
units on a scale | -3.2 (12.94)

ADVERSE EVENTS:
Time Frame: Up to 7 months
Arm/Group | Aripiprazole Lauroxil
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 5/51
Other Adverse Events (participants affected / at risk) | 3/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole Lauroxil (N=51)
Psychotic disorder (Psychiatric disorders) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole Lauroxil (N=51)
Anxiety (Psychiatric disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should an Investigator desire to disclose study results, Sponsor will review the results disclosure prior to public release and can embargo the disclosure for a period of at least 60 days. Revisions to the disclosure will be negotiated in good faith. For a multicenter study the Investigators agree to publish/publicly present the results together with the other sites for the 12 month period after study results are available unless Sponsor grants written permission in advance.

DOCUMENTS (2):
  • Study Protocol (2016-09-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT02634320/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-18): https://cdn.clinicaltrials.gov/large-docs/20/NCT02634320/SAP_001.pdf